CLINICAL TRIAL: NCT03589430
Title: Haemostatic Imbalance in Patients With Chronic Liver Disease- Its Relation to Severity and Outcome
Brief Title: Haemostatic Imbalance in Patients With Chronic Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mohammed Mahrous Sayed, principal investigator, Assiut University
Other Study IDs: Haemostasis imbalance in CLD
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Haemostasis Imbalance in Chronic Liver Disease
MeSH Terms: interventions — Protein C; Protein S; Antithrombin III

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1 child A: child A liver cirrhosis
  Interventions: Other: Laboratory investigations ( protein C, protein S , antithrombin III)
- 2 child B: child B liver cirrhosis
  Interventions: Other: Laboratory investigations ( protein C, protein S , antithrombin III)
- 3 child C: child C liver cirrhosis
  Interventions: Other: Laboratory investigations ( protein C, protein S , antithrombin III)

INTERVENTIONS:
Other: Laboratory investigations ( protein C, protein S , antithrombin III) — laboratory investigations ( protein C , protein S , antithrombin)

SUMMARY:
To assess the level of protein C, S ,antithrombin in patients with liver cirrhosis To correlate the level of these parameters with the degree of liver cirrhosis To correlate the level of procoagulants with the level of anticoagulant proteins in liver cirrhosis

DETAILED DESCRIPTION:
The liver has a cardinal role in the haemostatic system. Liver has the major role in synthesizing all clotting factors and coagulation inhibitors. Under the physiological conditions the balanced levels of procoagulant and anticoagulants determine the risk of hemorrhage and thrombosis.

In chronic liver disease due to chronic hepatitis and underlying cirrhosis, this haemostatic imbalance leads to hypercoagulability which favors thrombosis despite the longer coagulation times of their plasma, compared with that of healthy individuals. The end stage cirrhosis is however predominately associated with bleeding tendency.

Protein C (PC) and protein S (PS) are vitamin K-dependent glycoproteins, that act as natural anticoagulants.

Antithrombin III (AT III) is a natural anticoagulant that is synthesized exclusively in parenchymal cells of the liver The cause of hypercoagulability in chronic liver disease is the reduced level of protein C and increased level of factor VIIIa .As a consequence of hypercoagulability, the deep vein thrombosis, pulmonary embolism, hepatic and portal vein thrombosis may occur.

Varnika et al 2017 found a significantly low protein C value in both chronic hepatitis and cirrhosis group when compared with control group.

Acquired deficiency of АТ III can be caused by decreased synthesis due to damage to hepatic cells Patients with CLD were (and are still) subjected to laboratory screening with the prothrombin and activated partial thromboplastin times (PT and APTT), and those with abnormal values were (are) treated with plasma or procoagulant agents to correct the abnormalities and to prevent haemorrhage during invasive procedures or to stop bleeding from the gastrointestinal tract. Saja et al., and Saray et al 2009 found significantly low protein C value in both chronic hepatitis and cirrhosis group when compared with control group. This was a sign of reduced hepatocyte synthetic capacity in chronic hepatitis. Zocco et al 2009 showed that in CLD reduction in plasma levels of PC correlate with a higher Model For End-Stage Liver Disease (MELD) score. These findings, including the present one, confirm that levels of PC are sensitive markers .

Determination of the levels of AT III and aminotransferase activity in patients with liver disease may be used for differential diagnoses and the monitoring of disease progression.

Little attention had been paid to the fact that, similar to procoagulant factors, their anticoagulant counterparts (namely protein C [PC] and antithrombin) are also reduced to the same extent in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as liver cirrhosis confirmed clinical , biochemical and ultrasonography.
* severity of cirrhosis was assessed according to Child-Pugh score and MELD score.

Exclusion Criteria:

* history of bleeding or thrombotic disorder,
* history of renal disease, diabetes mellitus,
* ongoing or recent pregnancy,
* recent history of transfusion of blood products,
* current anticoagulation therapy.
* Hepatocellular carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Assesment of haemostatic profile in different stages of liver cirrhosis | baseline
  assessment of the level of protein C, S ,antithrombin in patients with liver cirrhosis, and correlate the level of these parameters with the degree of liver cirrhosis

SECONDARY OUTCOMES:
The value of anticoagulant use in patients with liver cirrhosis | baseline
  Cirrhotic patients has bleeding disorders and also high possibility of developing thrmobosis , so secondary to this study which assess the cause of hypercoaguability state in liver cirrhosis, new studies can be based on this study to assess the value of use of anticoagulant therapy in cirrhotic patients who are at high risk of developing thrombosis

REFERENCES:
- [Background] Rai V, Dhameja N, Kumar S, Shukla J, Singh R, Dixit VK. Haemostatic Profile of Patients with Chronic Liver Disease- its Correlation with Severity and Outcome. J Clin Diagn Res. 2017 Aug;11(8):EC24-EC26. doi: 10.7860/JCDR/2017/24975.10451. Epub 2017 Aug 1. PMID 28969137
- [Background] Wypasek E, Undas A. Protein C and protein S deficiency - practical diagnostic issues. Adv Clin Exp Med. 2013 Jul-Aug;22(4):459-67. PMID 23986205
- [Background] Hessien M, Ayad M, Ibrahim WM, ulArab BI. Monitoring coagulation proteins during progression of liver disease. Indian J Clin Biochem. 2015 Apr;30(2):210-6. doi: 10.1007/s12291-014-0429-1. Epub 2014 Apr 19. PMID 25883431
- [Background] Tripodi A, Anstee QM, Sogaard KK, Primignani M, Valla DC. Hypercoagulability in cirrhosis: causes and consequences. J Thromb Haemost. 2011 Sep;9(9):1713-23. doi: 10.1111/j.1538-7836.2011.04429.x. PMID 21729237